CLINICAL TRIAL: NCT02906319
Title: Association Between Serum 25-hydroxyvitamin D Levels and Glycated Haemoglobin in Diabetic Patients With Chronic Kidney Disease
Brief Title: Vitamin D and HbA1c Levels in Diabetic Patients With CKD
Status: Completed | Type: Observational
Sponsor: Ng Yong Muh (Other)
Collaborators: University of Malaya (Other); Malaysian Society of Nephrology (Unknown)
Responsible Party: Sponsor-Investigator, Ng Yong Muh, Dr, University of Malaya
Organization: University of Malaya (Other)
Other Study IDs: 201412-878
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Vitamin D Deficiency; Diabetes Mellitus
MeSH Terms: conditions — Vitamin D Deficiency; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the association between serum 25-hydroxyvitamin D and HbA1c levels in diabetic patients with chronic kidney disease. The investigators hypothesized that serum 25-hydroxyvitamin D levels were negatively correlated with HbA1c levels.

DETAILED DESCRIPTION:
This was a cross sectional study using consecutive sampling methodology for participant recruitment. It was carried out at the specialized diabetic, renal, and general outpatient clinics in the University of Malaya Medical Centre (UMMC), Kuala Lumpur, Malaysia.

Serum 25(OH)D levels were determined by using direct chemiluminesent immunoassay (ADVIA Centaur XP; Siemens Healthcare Diagnostics, Tarrytown, New York, USA). Serum HbA1c levels were determined using high-pressure liquid chromatography (Variant™ II Turbo; Bio-Rad, Hercules, California, USA).

Data collected will be analyzed using Statistical Package for Social Sciences SPSS version 23.0 for Windows, version 23.0 (IBM Corp., Armonk, New York, USA).

ELIGIBILITY:
Inclusion Criteria:

* eGFR 15-59 ml/min/1.73m2
* age ≥ 18 years old
* able to provide informed consent

Exclusion Criteria:

* active infections
* autoimmune diseases
* malignancies
* on immunosuppressive therapy
* on vitamin D supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who attended specialized diabetic, renal, and general outpatient clinics in the University of Malaya Medical Centre (UMMC), Kuala Lumpur, Malaysia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D levels | Within 2 weeks from enrolment
  The unit of measure was nmol/L. The detection limit of the device was <10 nmol/L. A mean value of 5 nmol/L were taken for results reported as <10nmol/L.
HbA1c levels | Within 2 weeks from enrolment
  The unit of measure was percentage (using NGSP standarization).

CONTACTS AND LOCATIONS:
Overall Officials: Yong Muh Ng, MMed, Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: Yes
A dataset of participants' clinical characteristics and biochemical tests result. The data was obtained directly from the participants and via Laboratory Information System. It is ready for submission.